CLINICAL TRIAL: NCT06831474
Title: Excretion of Rivaroxaban in Human Breast Milk
Acronym: LACT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Rupsa C. Boelig, Associate Professor, Thomas Jefferson University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: iRISID-2025-0397
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Postpartum; VTE Prophylaxis; VTE (Venous Thromboembolism); Rivaroxaban; Breastfeeding; Breast Milk Collection
Keywords: Rivaroxaban; Relative infant dose; LACT; Rivaroxaban in breast milk
MeSH Terms: conditions — Venous Thromboembolism; Breast Feeding; Breast Milk Expression | interventions — Rivaroxaban; Tablets

STUDY DESIGN:
Intervention Model Description: This is a prospective phase 1, two arm drug trial comparing the excretion of rivaroxaban in human breast milk between groups receiving prophylactic or therapeutic dosing during the postpartum period. Patients will be screened and enrolled for participation either antepartum or postpartum.
  Once postpartum, patients will be re-screened for any exclusion criteria and to be sure all inclusion criteria is met. Prior to receiving rivaroxaban each patient will provide a baseline 1 mL breast milk sample. Patients will either receive 10 mg or 20 mg daily of rivaroxaban starting by the first postpartum day. The dose will be be ordered by their postpartum physician team through the inpatient pharmacy and dispensed by their inpatient nursing team, as per standard of care at the discretion of their physician. 1 mL of breast milk will be collected at 3, 6, 12, 15 and 24 hours following their first morning dose. The patient will continue the medication while in house and for each subsequent day o
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Prophylactic rivaroxaban (Active Comparator): Patients will receive 10 mg daily of rivaroxaban starting by the first postpartum day. The medication will be ordered by their postpartum physician team through the inpatient pharmacy and dispensed by their inpatient nursing team, as per standard of care. The decision for dose 10 mg vs 20 mg of rivaroxaban is based on inclusion criteria and patient's physician team's recommendation for prophylactic (10 mg) vs. therapeutic (20 mg) dosing.
  Interventions: Drug: Rivaroxaban 10 MG Oral Tablet
- Therapeutic or Intermediate dose rivaroxaban (Active Comparator): Patients will receive 20 mg daily of rivaroxaban starting by the first postpartum day. The medication will be ordered by their postpartum physician team through the inpatient pharmacy and dispensed by their inpatient nursing team, as per standard of care. The decision for 10 mg vs 20 mg of rivaroxaban is based on inclusion criteria and patient's physician team's recommendation for prophylactic (10 mg) vs. therapeutic (20 mg) dosing.
  Interventions: Drug: Rivaroxaban 20 MG Oral Tablet

INTERVENTIONS:
Drug: Rivaroxaban 10 MG Oral Tablet — 10mg rivaroxaban daily
  Other Names: Xarelto
  Arms: Prophylactic rivaroxaban
Drug: Rivaroxaban 20 MG Oral Tablet — 20mg rivaroxaban daily
  Arms: Therapeutic or Intermediate dose rivaroxaban

SUMMARY:
The purpose of this study is to investigate the distribution of rivaroxaban into human milk at both therapeutic and prophylactic doses, and over time with repeated dosing.

DETAILED DESCRIPTION:
The aim of our study is to perform a phase 1, single arm clinical trial to investigate the distribution of rivaroxaban into human milk at both therapeutic and prophylactic maternal doses. Our goal is to enhance the limited, although positive, data regarding the safety of rivaroxaban in breastfeeding. Our novel contributions to the existing body of literature will be in our investigation of rivaroxaban at both prophylactic and therapeutic doses, in repeated doses over time, and in a larger sample of participants. These results will provide physicians and national societies with safety data needed to properly counsel patients and advance clinical guidelines for postpartum care.

ELIGIBILITY:
Inclusion Criteria:

1. Postpartum within 6 weeks of delivery
2. Greater than 18 years old at expected date of delivery
3. English speaking
4. Hemodynamically stable without concern for ongoing blood loss
5. Non-breastfeeding
6. Or breastfeeding an infant born at or equal to 37 weeks' gestation, weighing >2600g at birth and is not requiring intensive care
7. Meet inclusion criteria for prophylactic rivaroxaban dose: pre-pregnancy BMI >/= 40 and/or any personal history of VTE. Or >/= 2 of the following: pre-pregnancy BMI 30-39, immobility, pregnancy complications, cesarean delivery, hysterectomy
8. Or meet inclusion criteria for therapeutic rivaroxaban dose: have an indication for therapeutic anticoagulation per the American College of Obstetricians and Gynecologists' (ACOG) practice bulletin #196, or other indication per their primary team, and recommended for such anticoagulation per their primary practitioner.

Exclusion Criteria:

1. Pregnant
2. Less than 18 years old at estimated date of delivery
3. Hemodynamic instability and/or concern for ongoing blood loss
4. Newly diagnosed deep vein thrombosis (DVT) or pulmonary embolism (PE) in the postpartum period
5. Abnormal maternal renal or liver function (creatinine clearance < 30 mL/min and/or liver function tests greater than lab normal)
6. A contraindication to rivaroxaban: hypersensitivity to rivaroxaban; active pathological bleeding
7. Breastfeeding an infant admitted to neonatal intensive care unit, infant gestational age at birth <37w0d or weighing <2600g.
8. If all of the following are met: age less than 40, ambulating, body mass index (BMI) less than 30, no active history of malignancy.
9. If patient lacks indication for therapeutic anticoagulation in the postpartum period per the American College of Obstetricians and Gynecologists' (ACOG) practice bulletin #196

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of rivaroxaban in breast milk | Postpartum day 1
  Time/Concentration profile of rivaroxaban in breast milk prior to intake (0) and 3, 6, 12, 15 and 24 hours following morning dose on day 0-1
Concentration of rivaroxaban in breast milk | Postpartum week 6
  Time/concentration profile of rivaroxaban in breast milk 3 hours following morning dose on day 2 and onward
Absolute infant dose of rivaroxaban | 6 week postpartum
  The absolute infant dose is calculated from average drug concentrations in breast milk multiplied by an estimated breast milk intake of 150 mL/kg/day.
Relative infant dose | 6 weeks postpartum
  The relative infant dose is the absolute infant dose expressed as a percentage of the weight adjusted maternal dose, based on an average maternal weight of 75 kg. It is expressed in mg/kg/day.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The participant data will be kept confidential and access will be limited to the study investigators in order to respect the privacy of the participants.

REFERENCES:
- [Background] Male C, Lensing AWA, Palumbo JS, Kumar R, Nurmeev I, Hege K, Bonnet D, Connor P, Hooimeijer HL, Torres M, Chan AKC, Kenet G, Holzhauer S, Santamaria A, Amedro P, Chalmers E, Simioni P, Bhat RV, Yee DL, Lvova O, Beyer-Westendorf J, Biss TT, Martinelli I, Saracco P, Peters M, Kallay K, Gauger CA, Massicotte MP, Young G, Pap AF, Majumder M, Smith WT, Heubach JF, Berkowitz SD, Thelen K, Kubitza D, Crowther M, Prins MH, Monagle P; EINSTEIN-Jr Phase 3 Investigators. Rivaroxaban compared with standard anticoagulants for the treatment of acute venous thromboembolism in children: a randomised, controlled, phase 3 trial. Lancet Haematol. 2020 Jan;7(1):e18-e27. doi: 10.1016/S2352-3026(19)30219-4. Epub 2019 Nov 5. PMID 31699660
- [Background] Muysson M, Marshall K, Datta P, Rewers-Felkins K, Baker T, Hale TW. Rivaroxaban Treatment in Two Breastfeeding Mothers: A Case Series. Breastfeed Med. 2020 Jan;15(1):41-43. doi: 10.1089/bfm.2019.0124. Epub 2019 Sep 18. PMID 31532233
- [Background] Saito J, Kaneko K, Yakuwa N, Kawasaki H, Yamatani A, Murashima A. Rivaroxaban Concentration in Breast Milk During Breastfeeding: A Case Study. Breastfeed Med. 2019 Dec;14(10):748-751. doi: 10.1089/bfm.2019.0230. Epub 2019 Nov 20. PMID 31746638
- [Background] Wiesen MH, Blaich C, Muller C, Streichert T, Pfister R, Michels G. The Direct Factor Xa Inhibitor Rivaroxaban Passes Into Human Breast Milk. Chest. 2016 Jul;150(1):e1-4. doi: 10.1016/j.chest.2016.01.021. PMID 27396794
- [Background] Zhao Y, Arya R, Couchman L, Patel JP. Are apixaban and rivaroxaban distributed into human breast milk to clinically relevant concentrations? Blood. 2020 Oct 8;136(15):1783-1785. doi: 10.1182/blood.2020006231. No abstract available. PMID 32488251
- [Background] Bennett PN, ed. Drugs and human lactation, 2nd ed. Amsterdam. Elsevier. 1996.
- [Background] Lanitis T, Leipold R, Hamilton M, Rublee D, Quon P, Browne C, Cohen AT. Cost-effectiveness of Apixaban Versus Other Oral Anticoagulants for the Initial Treatment of Venous Thromboembolism and Prevention of Recurrence. Clin Ther. 2016 Mar;38(3):478-93.e1-16. doi: 10.1016/j.clinthera.2016.01.020. Epub 2016 Feb 26. PMID 26922297
- [Background] Guillonneau M, de Crepy A, Aufrant C, Hurtaud-Roux MF, Jacqz-Aigrain E. [Breast-feeding is possible in case of maternal treatment with enoxaparin]. Arch Pediatr. 1996 May;3(5):513-4. doi: 10.1016/0929-693x(96)86421-9. No abstract available. French. PMID 8763733
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics. ACOG Practice Bulletin No. 196: Thromboembolism in Pregnancy. Obstet Gynecol. 2018 Jul;132(1):e1-e17. doi: 10.1097/AOG.0000000000002706. PMID 29939938